CLINICAL TRIAL: NCT01590472
Title: Consortium for the Sharing of Germ Line DNA and Tissue From Subjects With Mesothelioma
Brief Title: Do Your Genes Put You at a Higher Risk of Developing Mesothelioma
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Collaborators: University of Pennsylvania (Other); Mayo Clinic (Other); NYU Langone Health (Other); Johns Hopkins University (Other); Memorial Sloan Kettering Cancer Center (Other); Mesothelioma Applied Research Foundation, Inc. (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: GTS 36076 MARF
Record Dates: First submitted 2012-04-23; First posted 2012-05-03 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-05

CONDITIONS: Mesothelioma
Keywords: Genetics of Mesothelioma; Mesothelioma Consortium; GWAS; Asbestos
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mesothelioma: Individuals who have been diagnosed with mesothelioma

SUMMARY:
The purpose of this research study is to investigate the possibility that a person's genes put a person at a higher risk of developing mesothelioma. The investigators will examine genes from DNA (genetic material) isolated from blood. This study will also examine the impact of environmental and work exposures and family history of common cancers on the development of mesothelioma. The genetic markers in this study will basically identify how a person's body processes frequently encountered environmental pollutants and will not tell about chromosomes, specific diseases, or other potential health problems.

DETAILED DESCRIPTION:
Mesothelioma is a cancer that develops from serosal surfaces usually in response to prior asbestos exposure. A history of asbestos exposure can be elicited in more than 80% of mesothelioma victims. However, asbestos exposure alone is not sufficient to cause the development of mesothelioma. Nearly 27 million individuals in the US, were exposed to asbestos in the work place between 1940 and 1979 but just 3,000 new cases of mesothelioma are diagnosed each year. Therefore, the investigators hypothesis is that genetic variation in addition to asbestos exposure, and host factors contribute to the development of mesothelioma. It is estimated, based on the investigators preliminary studies, that a population in excess of 1,000 subjects with mesothelioma is required to perform a valid GWAS.

Therefore a multicenter approach is necessary to collect data and DNA on sufficient numbers with mesothelioma to adequately evaluate genetic risk. It is the aim of this proposal to develop a consortium of mesothelioma investigators to share phenotypic data and DNA samples and to perform genome wide association scanning (GWAS).

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to provide informed consent who suffer from mesothelioma

Exclusion Criteria:

* Inability to provide informed consent
* Absence of mesothelioma in self

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the clinics and in patient wards of the academic medical centers noted as collaborators.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Creation of a consortium of investigators (6 sites) for collection of blood for germline DNA and demographic information from 1000 mesothelioma subjects. | Participants will be seen on one occasion lasting 30-60 min to draw blood and elicit demographic information. It will require up to 2 years to enroll 1000 subjects with mesothelioma from the various sites.
  Demographic variables that will be collected include; date of birth, gender, age at first exposure to asbestos, type of exposure (occupational or bystander), family health history, personal past medical history, smoking history, age at diagnosis, latency, tumor location and cell type.

SECONDARY OUTCOMES:
GWAS will be performed on the DNA from the 1000 subjects with mesothelioma and compared with 1000 age and asbestos exposure matched controls free of past personal history and family history of cancer. | It will take up to 1 year, after the collection of the 1000 mesothelioma samples, to perform and analyze the GWAS.
  Given the significant risk for cancers other than the index mesothelioma in both subjects and their 1st degree relative (nearly 3 fold for sibs, parents and the mesothelioma subjects themselves and 7 fold for their children), the goal is to identify SNPs involved with mesothelioma and other common cancer susceptibility.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ohar, MD, Study Director — Wake Forest University; Lee Krug, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Julie Brahmer, MD, Principal Investigator — Johns Hopkins University; Harvey I Pass, MD, Principal Investigator — NYU Langone Health; Tobias Peikert, MD, Principal Investigator — Mayo Clinic; Daniel H Sterman, MD, Principal Investigator — University of Pennsylvania
Locations (6):
- United States (6):
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - New York University School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Bertazzi PA. Descriptive epidemiology of malignant mesothelioma. Med Lav. 2005 Jul-Aug;96(4):287-303. PMID 16457426
- [Background] Paul S, Neragi-Miandoab S, Jaklitsch MT. Preoperative assessment and therapeutic options for patients with malignant pleural mesothelioma. Thorac Surg Clin. 2004 Nov;14(4):505-16, ix. doi: 10.1016/j.thorsurg.2004.06.008. PMID 15559057
- [Background] Xu L, Flynn BJ, Ungar S, Pass HI, Linnainmaa K, Mattson K, Gerwin BI. Asbestos induction of extended lifespan in normal human mesothelial cells: interindividual susceptibility and SV40 T antigen. Carcinogenesis. 1999 May;20(5):773-83. doi: 10.1093/carcin/20.5.773. PMID 10334193
- [Background] Bocchetta M, Di Resta I, Powers A, Fresco R, Tosolini A, Testa JR, Pass HI, Rizzo P, Carbone M. Human mesothelial cells are unusually susceptible to simian virus 40-mediated transformation and asbestos cocarcinogenicity. Proc Natl Acad Sci U S A. 2000 Aug 29;97(18):10214-9. doi: 10.1073/pnas.170207097. PMID 10954737
- [Background] Kamp DW, Weitzman SA. Asbestosis: clinical spectrum and pathogenic mechanisms. Proc Soc Exp Biol Med. 1997 Jan;214(1):12-26. doi: 10.3181/00379727-214-44065. PMID 9012357
- [Background] Sluis-Cremer GK. Asbestos disease at low exposures after long residence times. Ann N Y Acad Sci. 1991 Dec 31;643:182-93. doi: 10.1111/j.1749-6632.1991.tb24461.x. No abstract available. PMID 1809131
- [Background] Neragi-Miandoab S. Multimodality approach in management of malignant pleural mesothelioma. Eur J Cardiothorac Surg. 2006 Jan;29(1):14-9. doi: 10.1016/j.ejcts.2005.10.008. Epub 2005 Dec 15. PMID 16343925
- [Background] Berry G, Wagner JC. Effect of age at inoculation of asbestos on occurrence of mesotheliomas in rats. Int J Cancer. 1976 Apr 15;17(4):477-83. doi: 10.1002/ijc.2910170410. PMID 1279040
- [Background] Becklake MR, Toyota B, Stewart M, Hanson R, Hanley J. Lung structure as a risk factor in adverse pulmonary responses to asbestos exposure. A case-referent study in Quebec chrysotile miners and millers. Am Rev Respir Dis. 1983 Sep;128(3):385-8. doi: 10.1164/arrd.1983.128.3.385. PMID 6311060
- [Background] Spirtas R, Heineman EF, Bernstein L, Beebe GW, Keehn RJ, Stark A, Harlow BL, Benichou J. Malignant mesothelioma: attributable risk of asbestos exposure. Occup Environ Med. 1994 Dec;51(12):804-11. doi: 10.1136/oem.51.12.804. PMID 7849863
- [Background] Baris YI, Sahin AA, Ozesmi M, Kerse I, Ozen E, Kolacan B, Altinors M, Goktepeli A. An outbreak of pleural mesothelioma and chronic fibrosing pleurisy in the village of Karain/Urgup in Anatolia. Thorax. 1978 Apr;33(2):181-92. doi: 10.1136/thx.33.2.181. PMID 663877
- [Background] Baris I, Simonato L, Artvinli M, Pooley F, Saracci R, Skidmore J, Wagner C. Epidemiological and environmental evidence of the health effects of exposure to erionite fibres: a four-year study in the Cappadocian region of Turkey. Int J Cancer. 1987 Jan 15;39(1):10-7. doi: 10.1002/ijc.2910390104. PMID 3025107
- [Background] Amundadottir LT, Sulem P, Gudmundsson J, Helgason A, Baker A, Agnarsson BA, Sigurdsson A, Benediktsdottir KR, Cazier JB, Sainz J, Jakobsdottir M, Kostic J, Magnusdottir DN, Ghosh S, Agnarsson K, Birgisdottir B, Le Roux L, Olafsdottir A, Blondal T, Andresdottir M, Gretarsdottir OS, Bergthorsson JT, Gudbjartsson D, Gylfason A, Thorleifsson G, Manolescu A, Kristjansson K, Geirsson G, Isaksson H, Douglas J, Johansson JE, Balter K, Wiklund F, Montie JE, Yu X, Suarez BK, Ober C, Cooney KA, Gronberg H, Catalona WJ, Einarsson GV, Barkardottir RB, Gulcher JR, Kong A, Thorsteinsdottir U, Stefansson K. A common variant associated with prostate cancer in European and African populations. Nat Genet. 2006 Jun;38(6):652-8. doi: 10.1038/ng1808. Epub 2006 May 7. PMID 16682969
- [Background] Freedman ML, Haiman CA, Patterson N, McDonald GJ, Tandon A, Waliszewska A, Penney K, Steen RG, Ardlie K, John EM, Oakley-Girvan I, Whittemore AS, Cooney KA, Ingles SA, Altshuler D, Henderson BE, Reich D. Admixture mapping identifies 8q24 as a prostate cancer risk locus in African-American men. Proc Natl Acad Sci U S A. 2006 Sep 19;103(38):14068-73. doi: 10.1073/pnas.0605832103. Epub 2006 Aug 31. PMID 16945910
- [Background] Rai AJ, Flores RM, Mathew A, Gonzalez-Espinoza R, Bott M, Ladanyi M, Rusch V, Fleisher M. Soluble mesothelin related peptides (SMRP) and osteopontin as protein biomarkers for malignant mesothelioma: analytical validation of ELISA based assays and characterization at mRNA and protein levels. Clin Chem Lab Med. 2010 Feb;48(2):271-8. doi: 10.1515/CCLM.2010.066. PMID 20131968
- [Background] Tajima K, Ohashi R, Sekido Y, Hida T, Nara T, Hashimoto M, Iwakami S, Minakata K, Yae T, Takahashi F, Saya H, Takahashi K. Osteopontin-mediated enhanced hyaluronan binding induces multidrug resistance in mesothelioma cells. Oncogene. 2010 Apr 1;29(13):1941-51. doi: 10.1038/onc.2009.478. Epub 2010 Jan 18. PMID 20101228
- [Background] Ohashi R, Tajima K, Takahashi F, Cui R, Gu T, Shimizu K, Nishio K, Fukuoka K, Nakano T, Takahashi K. Osteopontin modulates malignant pleural mesothelioma cell functions in vitro. Anticancer Res. 2009 Jun;29(6):2205-14. PMID 19528482
- [Background] Cerhan JR, Ansell SM, Fredericksen ZS, Kay NE, Liebow M, Call TG, Dogan A, Cunningham JM, Wang AH, Liu-Mares W, Macon WR, Jelinek D, Witzig TE, Habermann TM, Slager SL. Genetic variation in 1253 immune and inflammation genes and risk of non-Hodgkin lymphoma. Blood. 2007 Dec 15;110(13):4455-63. doi: 10.1182/blood-2007-05-088682. Epub 2007 Sep 7. PMID 17827388
- [Background] Langsenlehner U, Renner W, Yazdani-Biuki B, Eder T, Wascher TC, Paulweber B, Clar H, Hofmann G, Samonigg H, Krippl P. Integrin alpha-2 and beta-3 gene polymorphisms and breast cancer risk. Breast Cancer Res Treat. 2006 May;97(1):67-72. doi: 10.1007/s10549-005-9089-4. PMID 16317580
- [Background] Gerger A, Hofmann G, Langsenlehner U, Renner W, Weitzer W, Wehrschutz M, Wascher T, Samonigg H, Krippl P. Integrin alpha-2 and beta-3 gene polymorphisms and colorectal cancer risk. Int J Colorectal Dis. 2009 Feb;24(2):159-63. doi: 10.1007/s00384-008-0587-9. Epub 2008 Oct 3. PMID 18836731
- [Background] O'Donnell CJ, Nabel EG. Cardiovascular genomics, personalized medicine, and the National Heart, Lung, and Blood Institute: part I: the beginning of an era. Circ Cardiovasc Genet. 2008 Oct;1(1):51-7. doi: 10.1161/CIRCGENETICS.108.813337. PMID 20031542
- [Background] Ohar J, Sterling DA, Bleecker E, Donohue J. Changing patterns in asbestos-induced lung disease. Chest. 2004 Feb;125(2):744-53. doi: 10.1378/chest.125.2.744. PMID 14769760
- [Background] Hirschhorn JN, Daly MJ. Genome-wide association studies for common diseases and complex traits. Nat Rev Genet. 2005 Feb;6(2):95-108. doi: 10.1038/nrg1521. PMID 15716906
- [Background] Boezen HM. Genome-wide association studies: what do they teach us about asthma and chronic obstructive pulmonary disease? Proc Am Thorac Soc. 2009 Dec;6(8):701-3. doi: 10.1513/pats.200907-058DP. PMID 20008879
- [Background] Landi S, Gemignani F, Neri M, Barale R, Bonassi S, Bottari F, Canessa PA, Canzian F, Ceppi M, Filiberti R, Ivaldi GP, Mencoboni M, Scaruffi P, Tonini GP, Mutti L, Puntoni R. Polymorphisms of glutathione-S-transferase M1 and manganese superoxide dismutase are associated with the risk of malignant pleural mesothelioma. Int J Cancer. 2007 Jun 15;120(12):2739-43. doi: 10.1002/ijc.22590. PMID 17290392
- [Background] Dianzani I, Gibello L, Biava A, Giordano M, Bertolotti M, Betti M, Ferrante D, Guarrera S, Betta GP, Mirabelli D, Matullo G, Magnani C. Polymorphisms in DNA repair genes as risk factors for asbestos-related malignant mesothelioma in a general population study. Mutat Res. 2006 Jul 25;599(1-2):124-34. doi: 10.1016/j.mrfmmm.2006.02.005. Epub 2006 Mar 27. PMID 16564556
- [Background] Robinson BW, Lake RA. Advances in malignant mesothelioma. N Engl J Med. 2005 Oct 13;353(15):1591-603. doi: 10.1056/NEJMra050152. No abstract available. PMID 16221782
- [Background] Robinson BW, Musk AW, Lake RA. Malignant mesothelioma. Lancet. 2005 Jul 30-Aug 5;366(9483):397-408. doi: 10.1016/S0140-6736(05)67025-0. PMID 16054941
- [Background] Wheatley-Price P, Yang B, Patsios D, Patel D, Ma C, Xu W, Leighl N, Feld R, Cho BC, O'Sullivan B, Roberts H, Tsao MS, Tammemagi M, Anraku M, Chen Z, de Perrot M, Liu G. Soluble mesothelin-related Peptide and osteopontin as markers of response in malignant mesothelioma. J Clin Oncol. 2010 Jul 10;28(20):3316-22. doi: 10.1200/JCO.2009.26.9944. Epub 2010 May 24. PMID 20498407
- [Background] Ohar JA, Ampleford EJ, Howard SE, Sterling DA. Identification of a mesothelioma phenotype. Respir Med. 2007 Mar;101(3):503-9. doi: 10.1016/j.rmed.2006.06.028. Epub 2006 Aug 21. PMID 16919927
- [Background] Gudmundsson J, Sulem P, Steinthorsdottir V, Bergthorsson JT, Thorleifsson G, Manolescu A, Rafnar T, Gudbjartsson D, Agnarsson BA, Baker A, Sigurdsson A, Benediktsdottir KR, Jakobsdottir M, Blondal T, Stacey SN, Helgason A, Gunnarsdottir S, Olafsdottir A, Kristinsson KT, Birgisdottir B, Ghosh S, Thorlacius S, Magnusdottir D, Stefansdottir G, Kristjansson K, Bagger Y, Wilensky RL, Reilly MP, Morris AD, Kimber CH, Adeyemo A, Chen Y, Zhou J, So WY, Tong PC, Ng MC, Hansen T, Andersen G, Borch-Johnsen K, Jorgensen T, Tres A, Fuertes F, Ruiz-Echarri M, Asin L, Saez B, van Boven E, Klaver S, Swinkels DW, Aben KK, Graif T, Cashy J, Suarez BK, van Vierssen Trip O, Frigge ML, Ober C, Hofker MH, Wijmenga C, Christiansen C, Rader DJ, Palmer CN, Rotimi C, Chan JC, Pedersen O, Sigurdsson G, Benediktsson R, Jonsson E, Einarsson GV, Mayordomo JI, Catalona WJ, Kiemeney LA, Barkardottir RB, Gulcher JR, Thorsteinsdottir U, Kong A, Stefansson K. Two variants on chromosome 17 confer prostate cancer risk, and the one in TCF2 protects against type 2 diabetes. Nat Genet. 2007 Aug;39(8):977-83. doi: 10.1038/ng2062. Epub 2007 Jul 1. PMID 17603485
- [Background] Gudmundsson J, Sulem P, Manolescu A, Amundadottir LT, Gudbjartsson D, Helgason A, Rafnar T, Bergthorsson JT, Agnarsson BA, Baker A, Sigurdsson A, Benediktsdottir KR, Jakobsdottir M, Xu J, Blondal T, Kostic J, Sun J, Ghosh S, Stacey SN, Mouy M, Saemundsdottir J, Backman VM, Kristjansson K, Tres A, Partin AW, Albers-Akkers MT, Godino-Ivan Marcos J, Walsh PC, Swinkels DW, Navarrete S, Isaacs SD, Aben KK, Graif T, Cashy J, Ruiz-Echarri M, Wiley KE, Suarez BK, Witjes JA, Frigge M, Ober C, Jonsson E, Einarsson GV, Mayordomo JI, Kiemeney LA, Isaacs WB, Catalona WJ, Barkardottir RB, Gulcher JR, Thorsteinsdottir U, Kong A, Stefansson K. Genome-wide association study identifies a second prostate cancer susceptibility variant at 8q24. Nat Genet. 2007 May;39(5):631-7. doi: 10.1038/ng1999. Epub 2007 Apr 1. PMID 17401366
- [Background] Smith DD. Women and mesothelioma. Chest. 2002 Dec;122(6):1885-6. doi: 10.1378/chest.122.6.1885. No abstract available. PMID 12475820
- [Background] Asbestos, asbestosis, and cancer: the Helsinki criteria for diagnosis and attribution. Scand J Work Environ Health. 1997 Aug;23(4):311-6. No abstract available. PMID 9322824
- [Background] Centers for Disease Control and Prevention (CDC). Malignant mesothelioma mortality--United States, 1999-2005. MMWR Morb Mortal Wkly Rep. 2009 Apr 24;58(15):393-6. PMID 19390506